CLINICAL TRIAL: NCT02071589
Title: Crossover Randomised Bioavailability Clinical Study Of A Single Dose Of Nifedipine Oral Solution From Laboratorio Reig Jofre S.A. Compared To Adalat(R) Capsules In Healthy Female Volunteers
Brief Title: Bioavailability Of A Single Dose Of Nifedipine Oral Solution Compared To Adalat Capsules In Healthy Female Volunteers
Acronym: NIFEPAR_PK1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reig Jofre Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2006-006159-11; CIM/06/300/04 (Other: CIM SANT PAU)
Record Dates: First submitted 2013-12-03; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine oral solution (Experimental): Nifedipine 5 mg/mL oral solution, 6 mL (30 mg of Nifedipine) at single dose
  Interventions: Drug: Nifedipine oral solution
- Nifedipine soft gelatine capsules (Active Comparator): Nifedipine soft gelatine capsules x3 (total 30 mg Nifedipine) at a single dose
  Interventions: Drug: Nifedipine soft gelatine capsules

INTERVENTIONS:
Drug: Nifedipine soft gelatine capsules — 3 Adalat capsules of 10 mg each one
  Other Names: Adalat
  Arms: Nifedipine soft gelatine capsules
Drug: Nifedipine oral solution — 6 mL of Nife Par solution
  Other Names: Nife-Par
  Arms: Nifedipine oral solution

SUMMARY:
Phase I, crossover, randomised, single dose, relative bioavailability clinical trial of a new oral solution of nifedipine compared to Adalat soft gelatine capsules in healthy female volunteers.

DETAILED DESCRIPTION:
The study was designed to compare the bioavailability of nifedipine new formulation specially designed to be used in pre-term labour management instead of anti-hypertensive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45.
* Body weight within the normal range (Quetelet index between 19 and 26) expressed as weight (kg) / height (m2) .
* Medical history , physical examination within normal appliances .
* No evidence of significant organic or psychiatric disease based on history, physical examination and laboratory tests .
* Laboratory tests (hematology and biochemistry) within the normal range , according to normal reference values of the Biochemistry laboratory of Hospital de la Santa Creu i Sant Pau. Variations may be allowed based on clinical judgment of the Centre d' Investigacio Medicament (CIM ) .
* Vital signs: blood pressure (Systolic Blood Pressure (SBP) > 90 <140 mm Hg / Diastolic Blood Pressure (DBP) > 50 <90 mm Hg ), heart rate (> 50 <90 ) , temperature and ECG record within normal range.
* Not having participated in another clinical trial during the previous three months at the beginning of the current study .
* Not having donated blood in the previous four weeks.
* Free acceptance to participate in the trial. Written informed consent signed.
* Use of effective contraception different from oral contraceptives.

Exclusion Criteria:

* Previous history of alcohol or drug use or abuse during the previous month to the selection process.
* High consumption of stimulant beverages (> 5 coffee, tea, cola drinks daily).
* Previous history of allergy, drug hypersensitivity or idiosyncrasy.
* Taking any medication in the 4 weeks preceding the trial, including non-prescription medicines and herbal remedies.
* Positive serology for hepatitis B, C or HIV.
* History or clinical evidence of cardiovascular disease, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological or other chronic diseases.
* Having had surgery during the previous 6 months.
* Having donated blood in the month before the study began.
* Smokers.
* Positive pregnancy test at any monitoring during the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-24h) | pre-dose and +10', +20', +30', +45', +1h, +1h15', +1h30', +2h, +3h, +5h, +7h, +9h, +12h y +24h post dose
Maximal plasmatic concentrations, Cmax | pre-dose and +10', +20', +30', +45', +1h, +1h15', +1h30', +2h, +3h, +5h, +7h, +9h, +12h y +24h post dose

SECONDARY OUTCOMES:
Time to maximal plasmatic concentrations, Tmax | pre-dose and +10', +20', +30', +45', +1h, +1h15', +1h30', +2h, +3h, +5h, +7h, +9h, +12h y +24h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Antonijoan, MD, PhD, Principal Investigator — CIM Sant Pau
Locations (1):
- CIM Sant Pau, Barcelona, Barcelona, Spain